CLINICAL TRIAL: NCT00620581
Title: Luteal Phase Administration of Paroxetine for the Treatment of PMDD: A Randomized, Double-Blind, Placebo-Controlled Trial in Canadian Women
Brief Title: Luteal Phase Administration of Paroxetine for the Treatment of PMDD
Acronym: PMDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Other Study IDs: BRL29060/621
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2005-11

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Paroxetine

ARMS (1):
- Paroxetine 10mg;paroxetine 20mg; Placebo (Placebo Comparator)
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — Paroxetine 10mg and 20mg during the luteal phase of the menstrual cycle

SUMMARY:
The efficacy of SSRI use to relieve the symptoms associated with premenstrual dysphoric disorder has been established. We proposed to test the hypothesis that intermittent treatment with paroxetine administered during the luteal phase of the menstrual cycle only is more effective than placebo in improving symptoms of PMDD. This was a double-blind, placebo-controlled, three-arm parallel group study of patients with PMDD. Menstruating women 18 years of age or older who met criteria for inclusion in the study were randomized to one of three arms: paroxetine 10mg/day during the luteal phase of the menstrual cycle; paroxetine 20mg/day during the luteal phase of the menstrual cycle; placebo daily during the luteal phase of the menstrual cycle. The objective was to evaluate the efficacy and safety of intermittent treatment of paroxetine in women with PMDD.

ELIGIBILITY:
Inclusion Criteria:

* PMDD according to DSM-IV criteria

Exclusion Criteria:

* Women were excluded if they were taking oral contraception, breast-feeding, pregnant, or planning to become pregnant during the study period.
* Women were also excluded if they met DSM-IV criteria for any Axis I disorder, were deemed a suicidal risk, had a history of SSRI use for premenstrual symptoms, were taking ongoing medication that could affect PMDD symptoms, had a clinically significant abnormality on screening blood tests, or had a baseline Montgomery-Asberg Depression Rating Scale score of equal to or greater than 10 during the follicular phase of the menstrual cycle.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Visual Analogue Scales

SECONDARY OUTCOMES:
PMTS-O; CGI-S; Sheehan Disability Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Concerns Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Steiner M, Ravindran AV, LeMelledo JM, Carter D, Huang JO, Anonychuk AM, Simpson SD. Luteal phase administration of paroxetine for the treatment of premenstrual dysphoric disorder: a randomized, double-blind, placebo-controlled trial in Canadian women. J Clin Psychiatry. 2008 Jun;69(6):991-8. doi: 10.4088/jcp.v69n0616. PMID 18517289